CLINICAL TRIAL: NCT02453022
Title: A Single Centre, Open-label, 5-Period, Cross Over, Randomized Study in Healthy Elderly Subjects to Evaluate the Relative Bioavailability of Hydrobromide Salt and Free Base Immediate Release Tablet Formulations of Danirixin in the Fed State, and to Evaluate the Effect of Food and Gastric Acid Secretion Suppression on Danirixin Pharmacokinetics Following Administration of Hydrobromide Salt Tablets
Brief Title: A 5-Period, Single Dose, Phase 1 Study in Healthy Elderly Subjects to Assess Relative Bioavailability and Food Effect of Two Oral Formulations of GSK1325756 (Free Base vs HBr Salt) and Food Effect on the HBr Formulation When Given With Omeprazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 201037
Record Dates: First submitted 2015-05-21; First posted 2015-05-25 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Bioavailability; Omeprazole; Danirixin; Food Effect; Pharmacokinetics
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Danirixin HBr + Danirixin FB + Omeprazole (Experimental): Subjects will receive danirixin FB 50 milligram (mg) immediate release (IR) tablet, single dose, in the fed state (treatment A), danirixin HBr 50 mg IR tablet, single dose, in the fed state (treatment B), danirixin HBr 50 mg IR tablet, single dose, in the fasted state (treatment C), or danirixin HBr 50 mg IR tablet, single dose, in the fed state (treatment D) as per randomization in period 1 to 4. In treatment Period 5, subjects will receive danirixin HBr 50 mg IR table, single dose, in the fed state with concomitant, steady state OMP (40 mg once daily for 5 days) (treatment E). Subject will receive treatment with washout period of 5 days in one of the four sequence DCABE, ADBCE, BACDE, CBDAE.
  Interventions: Drug: Danirixin HBr 50 mg IR Tablet; Drug: Danirixin FB 50 mg IR Tablet; Drug: Prilosec (omeprazole) 40mg Delayed-Release capsule

INTERVENTIONS:
Drug: Danirixin HBr 50 mg IR Tablet — Danirixin HBr 50 mg IR Tablet is white, film-coated, oval-shaped tablet for oral administration.
Drug: Danirixin FB 50 mg IR Tablet — Danirixin FB 50 mg IR Tablet is white, film-coated, capsule-shaped tablet for oral administration.
Drug: Prilosec (omeprazole) 40mg Delayed-Release capsule — Prilosec (omeprazole) 40 mg delayed-release capsule is opaque, hard gelatin, apricot, and amethyst colored capsules, coded 743 on cap and PRILOSEC 40 on the body for oral administration.

SUMMARY:
The current study will help to increase our understanding of the pharmacokinetics (PK) of danirixin. The primary objective of the study is to estimate the relative bioavailability of danirixin Hydrobromide (HBr) tablet, when compared to danirixin free base (FB). Safety and tolerability information for oral administration of danrixin HBr tablets in elderly subjects will also be obtained. Secondarily, this study will evaluate effect of food on PK of danirixin HBr, effect of gastric acid suppression, and within-subject PK variability of danirixin HBr. The outcome of this study will contribute to the selection of the most appropriate formulation/dosing regimen for future studies.

This is an open-label, 5-period crossover study. Study will be conducted in 18 healthy elderly subjects. Screening will occur within 42 days prior to Day 1 of period 1. The Treatment Periods will be separated by a washout period of a minimum 5 days. Follow-up will be done within 3 to 10 days post last dose.

ELIGIBILITY:
Inclusion Criteria:

* Between 65 and 80 years of age at screening (inclusive)
* Healthy, as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring or a subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included if the investigator and the GlaxoSmithKline (GSK) Medical Monitor agree that the finding is unlikely to introduce risk factors and will not interfere with the study procedures and objectives.
* Body Mass Index between 19 and 34 (inclusive)
* Male or Female Males: Male subjects with female partners of child bearing potential must comply with the following contraception requirements from the time of first dose of study medication until a cycle of spermatogenesis following five terminal half- lives after the last dose of study medication. a. Vasectomy with documentation of azoospermia. b. Male condom plus partner use of one of the contraceptive options: Contraceptive subdermal implant, Intrauterine device or intrauterine system, Oral Contraceptive, either combined or progestogen alone Injectable progestogen, Contraceptive vaginal ring, Percutaneous contraceptive patches.

This is an all-inclusive list of those methods that meet the following GSK definition of highly effective: having a failure rate of less than 1% per year when used consistently and correctly and, when applicable, in accordance with the product label. For non-product methods (e.g., male sterility), the investigator determines what is consistent and correct use. The GSK definition is based on the definition provided by the International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH). The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.

Females: A female subject is eligible to participate if she is not pregnant (as confirmed by a negative urine human chorionic gonadotrophin [hCG] test), not lactating, and at least one of the following conditions applies: Non-reproductive potential defined as: a. Pre-menopausal females with one of the following: Documented tubal ligation, Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, Hysterectomy, Documented Bilateral Oophorectomy. b. Postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause (refer to laboratory reference ranges for confirmatory levels)]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in protocol.
* Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin <= 1.5 × Upper limit of normal (ULN) (isolated bilirubin > 1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%).
* Resting Blood pressure (BP) of <=160/90 millimetre (mm) mercury (Hg), irrespective of anti-hypertensive medication status for the subject.
* Able to consume the Food and Drug Administration (FDA) defined high fat meal within 30 minutes in each of the four treatment periods where study treatment is administered in a fed state

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study Hepatitis B surface antigen (HBsAg) or positive Hepatitis C antibody (HCV Ab) result within 3 months of screening.
* A positive pre-study drug/alcohol screen, with the exception of a positive result considered by the investigator to be directly attributable to prescription medication approved for subject use during the study.
* A positive test for human immunodeficiency virus (HIV) antibody.
* Use of prescription or non-prescription drugs, including proton pump inhibitors, histamine receptor 2 antagonists, systemic antacid medications (unless these can be held during the study), vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study treatment until completion of the last study assessment for Period 5, unless in the opinion of the investigator and GSK Medical Monitor, the medication will not interfere with the study procedures or compromise subject safety. Some examples of exceptions (permitted medications) are: a. Stable dose of anti-hypertensive medication for at least 3 months prior to the screening visit. b. Stable dose of lipid-lowering medications (statins or fibrates) for at least 3 months prior to the screening visit. c. Antacids up to 24 hours prior to dosing This list is not meant to be all inclusive.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 3 months, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities (any investigational, non-marketed, non-FDA-approved medicine) within 12 months prior to the first dosing day.
* History of regular alcohol consumption within 6 months of the study defined as:

An average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 gram (g) of alcohol: a half-pint (approximately 240 millilitre [mL]) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.

* Urine cotinine levels indicative of current smoking, or history or regular use of tobacco- or nicotine-containing products, including e-cigarettes and nicotine patches, within 90 days prior to screening.
* Consumption of red wine, Seville oranges, grapefruit or grapefruit juice and/or pummelos, citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study treatment until collection of the final blood sample.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 3-month period.
* Unwillingness or inability to follow all of the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* Direct involvement in the conduct of the study, or relative of any person directly involved in the conduct of the study.
* Female Subjects: Positive urine beta-hCG test at screening.
* Screening QT interval corrected for heart rate according to Fridericia's formula (QTcF)> 450 millisecond (msec) or an ECG that is not suitable for QT measurements (e.g., poorly defined termination of T-wave).
* History of sensitivity to any of the study treatments, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-05-18 (Actual); Primary Completion 2015-07-31 (Actual); Study Completion 2015-07-31 (Actual)

PRIMARY OUTCOMES:
Composite of Danirixin PK parameters | Blood samples for PK analysis will be collected at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours (hrs) post-dose in each period
  Danirixin PK parameters area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC[0-inf]) and maximum observed concentration (Cmax) following single dose administration of FB tablet (reference), relative to HBr tablet (test) will be assessed.
Number of participants with adverse events (AE) /serious adverse event (SAE) as a measure of safety and tolerability | Up to Day 36
  AE/SAE will be collected from the start of study treatment and until the follow-up visit or contact for study treatment period 5. Intensity of AEs will be categorized as mild, moderate or severe. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity is a congenital anomaly/birth defect is associated with liver injury and impaired liver function.
Composite of vital signs as a measure of safety and tolerability | Up to Day 31
  Vital signs will include temperature, systolic and diastolic blood pressure, pulse rate, and respiratory rate.
Electrocardiogram (ECG) as a measure of safety and tolerability | Up to Day 29
  ECG will be obtained at selected time-points during the study.
Composite of clinical laboratory tests as a measure of safety and tolerability | Up to Day 31
  Clinical laboratory tests will include hematology, clinical chemistry and urinalysis.

SECONDARY OUTCOMES:
Composite of other Danirixin PK parameters | Blood samples for PK analysis will be collected at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 hrs post-dose in each period
  Other Danirixin PK parameters area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration within a subject across all treatments (AUC[0-t]), time of occurrence of Cmax (tmax), terminal phase half-life (t1/2), time of last quantifiable concentration (tlast) and lag time before observation of drug concentrations in sampled matrix (tlag) following single dose administration of FB tablet (reference), relative to HBr tablet (test) will be assessed.
Composite of Danirixin PK parameters to estimate the food effect | Blood samples for PK analysis will be collected at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 hrs post-dose in each period
  Danirixin PK parameters AUC(0-inf), AUC(0-t), Cmax, tmax, t1/2, tlast and tlag following danirixin HBr tablet formulation under fasting and fed state will be assessed.
Composite of Danirixin PK parameters to estimate the effect of Omepazole (OMP) | Blood samples for PK analysis will be collected at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 hrs post-dose in each period
  Danirixin PK parameters AUC(0-inf), AUC(0-t), Cmax, tmax, t1/2, tlast and tlag following danirixin HBr tablet formulation with or without concomitant, steady state OMP will be assessed.
Composite of Danirixin PK parameters to estimate the within-subject variability of danirixin | Blood samples for PK analysis will be collected at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 hrs post-dose in each period
  Danirixin PK parameters AUC(0-inf), AUC(0-t), Cmax following danirixin HBr tablet formulation under fed conditions will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- See also: Results for study 201037 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/201037?search=study&b'search_terms=201037'#rs